CLINICAL TRIAL: NCT00980551
Title: A Pilot Study of Intravenous Topotecan and Vincristine in Combination With Subconjunctival Carboplatin for Patients With a History of Bilateral Retinoblastoma and Refractory/Recurrent Intraocular Disease (IND# 104,942)
Brief Title: Pilot Study of Topotecan/Vincristine With Subconjunctival Carboplatin for Patients With Bilateral Retinoblastoma
Acronym: RELRB1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment and competing studies
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RELRB1
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Carboplatin; Topotecan; Vincristine; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topotecan/Vincristine with subtenon Carboplatin (Experimental)
  Interventions: Drug: subtenon Carboplatin; Drug: Topotecan Hydrochloride; Drug: Vincristine; Drug: Filgrastim

INTERVENTIONS:
Drug: subtenon Carboplatin — Available in 50mg, 150mg, 450 mg, 600mg vials. It is provided as a premixed aqueous solution or lyophilized powder for injection given on day 1/week 10 (cycles 1-3).
  Other Names: Paraplatin
Drug: Topotecan Hydrochloride — Each vial contains topotecan hydrochloride equivalent to 4 mg of topotecan as free base. Given intravenously on days 1-5 of each week (cycles 1-6).
  Other Names: Hycamtin
Drug: Vincristine — Each vial contains vincristine sulfate, 1 mg; mannitol, 100 mg; sterile water for injection; Acetic acid and sodium acetate are added for pH control. Given intravenously on day 1/week 1 (cycles 1-6).
  Other Names: Oncovin
Drug: Filgrastim — Supplied as a clear solution in 300 mcg/ml 1 ml or 1.6 ml vials and prefilled syringes containing 300mcg/0.5mL or 480mcg/0.8mL. Given intravenously on day 6 of each week (cycles 1-6).
  Other Names: Neupogen

SUMMARY:
The investigators are testing subtenon carboplatin in combination with vincristine and topotecan given by vein in the hopes of finding a drug combination that may be effective against retinoblastoma that has come back (recurrent) or is resistant to other treatment (refractory).

The goals of this study are:

* To decide if the drug combination is a useful treatment for recurrent or refractory retinoblastoma
* To test the safety of the drug combination and to see what kind of effects (good and bad) can be expected from the drug combination
* To measure visual changes before and after the study therapy
* To use a special MRI scan to measure brain function involved in vision processing, both before and after the study therapy

In this study, the investigators are also testing a new experimental way of giving carboplatin "subtenon carboplatin". The carboplatin will be given directly in the eye through a needle placed under the covering of the eye. This is to try to get more carboplatin to the retinoblastoma inside the eye.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≤ 10 years of age
* Diagnosis: Patients must have a history of bilateral Retinoblastoma AND Recurrent/Refractory Intra-Ocular Retinoblastoma considered not amenable to cure with local therapies alone (photocoagulation with argon laser, cryotherapy, transpupillary thermotherapy, radioactive plaque therapy).
* Therapeutic Options: Patient's disease status is one for which there are no known options proven to provide a high chance for ocular salvage or cure other than external beam radiation or enucleation.
* Remaining visual function in target eye (s) is required
* Life Expectancy of > 8 weeks
* Lansky ≥ 50
* Prior Therapy: Patients must have local relapsed/refractory disease after receiving standard upfront therapy involving at least one chemotherapeutic regimen. There is no limit to prior chemotherapeutic regimens permitted. Patients may have received previous intravenous carboplatin, but may not have received prior subtenon carboplatin or intravenous topotecan.
* Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study, as described below:

  * Myelosuppressive chemotherapy: patients must not have received myelosuppressive chemotherapy within 3 weeks of study enrollment
  * Biologic therapies: Patients must not have received biologic anti-cancer agents within one week of study enrollment
* Radiation therapy: Four weeks must have elapsed since external beam radiation therapy, if given.
* Adequate Bone Marrow Function Defined as:

  * Peripheral absolute neutrophil count (ANC) ≥ 750/µL
  * Platelet count ≥ 75,000/µL (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to enrollment)
  * Hemoglobin ≥ 8.0 gm/dL (may receive RBC transfusions)
* Adequate Renal Function Defined as:

  * Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 OR threshold creatinine values based on age/gender derived from the Schwartz formula for estimating GFR
* Adequate Liver Function Defined As:

  * Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
  * SGPT (ALT) ≤ 5 x upper limit of normal (ULN) for age
  * Serum albumin ≥ 2 g/dL

Exclusion Criteria:

* Extra-ocular retinoblastoma
* Asynchronous involvement of the contralateral eye, previously untreated
* Uncontrolled infection at time of protocol entry
* Concomitant Medications:

  * Growth factors that support platelet or white cell number or function must not have been administered within the past 3 days
  * Patients who are currently receiving investigational drugs, or who have received an investigational drug within the last 7 days, are ineligible
  * Patients who are currently receiving other anti-cancer agents are ineligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To estimate the event-free survival, where an event is defined at the ocular level as the need for non-protocol therapy defined as additional non-protocol chemotherapy, external beam radiation, or enucleation. | at 1 year
To estimate the patterns of response, and response rate of locally refractory retinoblastoma to combination intravenous and peri-ocular chemotherapy. | at 1 yr

SECONDARY OUTCOMES:
To describe the toxicities associated with the proposed regimen. | at 1 yr
To describe the histologic findings in the eyes ultimately requiring enucleation. | at 1 yr
To describe the visual acuity of patients with advanced intraocular retinoblastoma before and after the proposed therapy. | at 1 yr
To describe primary visual cortex function in patients with retinoblastoma via functional Magnetic Resonance Imaging (fMRI) technique both before and after the proposed therapy. | at 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: James Geller, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States